CLINICAL TRIAL: NCT07373080
Title: Hybrid Type-2 Effectiveness-Implementation Study of Brief Culturally Adapted Behavioral Activation Therapy Delivered by Primary Care Psychologists for Adults With Depression in Rural Indonesian Primary Care Setting: A Study Protocol of Pragmatic Parallel Cluster Randomized Controlled Trial
Brief Title: Brief Culturally Adapted Behavioral Activation Therapy for Adults With Depression in Rural Indonesian Primary Care: A Type-2 Hybrid Effectiveness-Implementation Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Salma Salma, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3415/UN1/PS.1/SD/PT.01.04/2025
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Depression in Adults
Keywords: depression; behavioral activation therapy; culturally adapted treatment; implementation science; hybrid trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Two-arms parallel cluster randomized controlled trial, hybrid effectiveness-implementation trial type-2 with mixed method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT Implementation Arm (Experimental): Twelve primary health centers will be randomized into BAT implementation arm or TAU arm equally. Six selected primary care psychologists from six primary health centers will receive 4-session online training and 2-session booster training on BAT as well as synchronous (biweekly) and asynchronous (throughout implementation) online supervision from local and international experts. Forty-eight participants (adult patients) from six primary health centers will receive individual face-to-face Brief Culturally Adapted Behavioral Activation Therapy (3 sessions).
  Interventions: Other: Training and supervisionon BAT
- TAU (Treatment-as-usual) (No Intervention): Six primary health centers will be grouped into control arm using online randomizer. No implementation strategy applied for these clusters. Forty-eight participants (adult patients) from six primary health centers will receive treatment-as-usual for depression from primary care psychologist with no restriction on intervention approach and number of sessions.

INTERVENTIONS:
Other: Training and supervisionon BAT — Implementation strategy: Training and Supervision
  Training: Primary care psychologists will receive training which consists of 4-session online training of Behavioral Activation Therapy (BAT), 2-session of booster training focusing on BA principle and therapy protocol, and clinical practice with 2 participants during pilot study. Four-session online training, 1 booster session, and clinical practice with 2 participants have been delivered during pilot study phase.
  Supervision: Supervision will be provided during BAT implementation in two forms: 1) biweekly synchronous online supervision, starting from week 3 after the first day of recruitment and 2) asynchronous online supervision through online shared spreadsheet, available throughout BAT implementation.
  Participants in BAT implementation arm will receive 3 individual face-to-face sessions of Brief Culturally Adapted Behavioral Activation Therapy.
  Arms: BAT Implementation Arm

SUMMARY:
This is a type-2 hybrid effectiveness-implementation study of brief culturally adapted behavioral activation for adults with depression in primary care setting. This clinical trial has two parallel aims: 1) to understand if brief culturally adapted behavioral activation therapy delivered by psychologist in primary care in individual face-to-face session is effective to reduce depressive symptoms among adult patients in Primary Healthcare Centers and 2) to test the outcome of clinical training and supervision on acceptability, feasibility, appropriateness, and fidelity of implementation of brief culturally adapted behavioral activation therapy in Primary Healthcare Centers. The main questions it aims to answer is:

1) Is brief culturally adapted behavioral activation intervention delivered by primary care psychologist effective in reducing depressive symptoms among adult patients with depression in primary care settings and 2) Are training and supervision effective in enhancing acceptability, feasibility, appropriateness and fidelity of implementation of brief culturally adapted behavioral activation therapy for adults with depression in primary care settings?

DETAILED DESCRIPTION:
Depression is among global burden of diseases with higher treatment gap in lower- and middle-income countries (LMICs), including Indonesia. Integrating mental health care into primary care is one of recommended strategy to close the treatment gap in LMICs and there has been such integration through the placement of primary care psychologist in one of rural districts in Indonesia. In the other hand, behavioral activation therapy (BAT) is a culturally adaptable evidence-based therapy for adults with depression. However, little is known about implementation strategy to enhance the adoption of BAT as well as its clinical effectiveness in Indonesian primary care.

This study aims to: 1) test clinical effectiveness of BAT with prior systematic cultural adaptation in reducing depressive symptoms among adults with depression in primary care and 2) test the effect of implementation strategies (i.e., training and supervision) on implementation outcomes (i.e., acceptability, feasibility, appropriateness, and fidelity). The results of this study will inform further study to scale up BAT implementation in Indonesian primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old
* scored 10 or above on PHQ-9
* provide informed consent

Exclusion Criteria:

* having diagnosis of bipolar disorder, psychotic disorders, or substance use disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Depressive Symptoms as Assessed by Patient Health Questionnaire-9 (PHQ-9) at 1 Week after Intervention | Baseline and 1 week post intervention
  Participants will fill the PHQ-9 as self-reported questionnaire using paper and pencil format, administered by research assistant. PHQ-9 consists of nine items with four response from 'not at all' (0) to 'nearly every day' (3). The score of the PHQ-9 ranges from 0 to 27 with higher score indicating higher depressive symptoms.
Participant's Acceptability of Intervention as Assessed by Client Satisfaction Questionnaire-8 (CSQ-8) | Post intervention (immediately after intervention completed)
  Acceptability is defined as the participant's perception that a given treatment is agreeable, palatable, or satisfactory and will be measured using CSQ-8. CSQ-8 consists of 8 items with four optional responses. The score of the questionnaire will range from 1 to 32 with higher score indicating acceptability of intervention.
Clinical Provider's Perceived Acceptability as Assessed by Acceptability of Intervention Measure (AIM) | through study completion, an average of 3 months
  Acceptability is defined as the clinical provider's perception that a given treatment is agreeable, palatable, or satisfactory and will be measured by Acceptability of Intervention Measure (AIM). AIM consists of four items with five Likert-based responses. The score of the scale will range from 1 to 20 with higher score indicating higher acceptability to the intervention.
Clinical Provider's Perceived Feasibility as Assessed by Feasibility of Intervention Measure (FIM) | through study completion, an average of 3 months
  Feasibility is defined as the perceived extent to which the intervention can be successfully used or carried out in primary care setting from participants and clinical providers' perspectives and will be measured by Feasibility of Intervention Measure (FIM). FIM consists of four items with five Likert-type responses. The score of the scale will range from 1 to 20 with higher score indicating higher feasibility of the intervention.
Clinical Provider's Perceived Appropriateness as Assessed by Intervention Appropriateness Measure (IAM) | through study completion, an average of 3 months
  Appropriateness is defined as the perceived fit, relevance, or compatibility of brief culturally adapted behavioral activation for adults with depression in primary care setting from participant's and clinical provider's perspectives, and measured by Intervention Appropriateness Measure (IAM). IAM consists of four items with five Likert-based responses. The score of the scale will range from 1 to 20 with higher score indicating higher appropriateness of the intervention.
Qualitative Feedback on Acceptability, Feasibility, and Appropriateness from Participants and Clinical Providers as Assessed using Semi-structured Interview | From enrollment to 1 week after intervention completed (for participants) through study completion, an average of 3 months (for clinical providers)
  Participants and clinical providers will be asked about their experiences in receiving or providing the intervention through individual qualitative interview to understand their perceived acceptability, feasibility, and appropriateness in a more detailed and comprehensive way.

SECONDARY OUTCOMES:
Rate of Remission or Recovery of Depression Diagnosis as Assessed by Structured Clinical Interview for DSM-5 (SCID-5) at 1 Week after Intervention | Post-intervention (1 week after intervention completed)
  Rate of remission or recovery will be calculated in percentage based on result of SCID-5 interview, administered by primary care psychologist. The result of clinical interview will categorize the participants into active depression or in remission or no diagnosis (fully recovered).
Change in Quality of Life from Baseline as Assessed by WHO Quality of Life Brief Version (WHOQOL-BREF) at 1 Week after Intervention | Baseline (week 0) and post-intervention (1 week after intervention completed)
  Participants will fill the WHOQOL-BREV as self-reported questionnaire using paper and pencil format, administered by research assistant. WHOQOL-BREV consists of 26 items with score on each item ranges from 0 to 5. The scale will produce quality of life profile which consists of overall perception of individual's quality of life, overall perception of individual's health, and four quality of life domains (physical health, psychological, social relationship, and environment). The score is calculated using mean score of each domain, then transformed to 4-20. Higher score of the domain indicates higher quality of life.
Change from Baseline in Anxiety as Assessed by Generalized Anxiety Disorder-7 (GAD-7) at 1 Week after Intervention | Baseline (week 0) and post-intervention (1 week after intervention completed)
  Anxiety is measured using Generalized Anxiety Disorder-7 (GAD-7) as a self-reported questionnaire using paper and pencil format, administered by research assistant. GAD-7 consists of seven items with four response on each item ranging from 0 to 4. The score of GAD-7 will range from 0 to 21 with higher score indicating higher anxiety.
Rate of Remission or Recovery in Depression Diagnosis 1-month after Intervention as Assessed by Structured Clinical Interview for DSM-5 (SCID-5) | One month after intervention
  Rate of remission or recovery will be calculated in percentage based on result of SCID-5 interview, administered by primary care psychologist. The result of clinical interview will categorize the participants into active depression or in remission or no diagnosis (fully recovered).
Change in Depressive Symptoms 1-month after Intervention as Assessed by Patient Health Questionnaire-9 (PHQ-9) | Baseline (week 0) and 1-month after intervention
  Participants will fill the PHQ-9 as self-reported questionnaire using paper and pencil format, administered by research assistant. PHQ-9 consists of nine items with four response from 'not at all' (0) to 'nearly every day' (3). The score of the PHQ-9 ranges from 0 to 27 with higher score indicating higher depressive symptoms.
Change in Quality of Life 1-month after Intervention as Assessed by WHO Quality of Life Brief Version (WHOQOL-BREF) | Baseline (week 0) and 1-month after intervention
  Participants will fill the WHOQOL-BREV as self-reported questionnaire using paper and pencil format, administered by research assistant. WHOQOL-BREV consists of 26 items with score on each item ranges from 0 to 5. The scale will produce quality of life profile which consists of overall perception of individual's quality of life, overall perception of individual's health, and four quality of life domains (physical health, psychological, social relationship, and environment). The score is calculated using mean score of each domain, then transformed to 4-20. Higher score of the domain indicates higher quality of life.
Change in Anxiety 1-month after Intervention as Assessed by Generalized Anxiety Disorder-7 (GAD-7) | Baseline (week 0) and 1-month after intervention
  Anxiety is measured using Generalized Anxiety Disorder-7 (GAD-7) as a self-reported questionnaire using paper and pencil format, administered by research assistant. GAD-7 consists of seven items with four response on each item ranging from 0 to 4. The score of GAD-7 will range from 0 to 21 with higher score indicating higher anxiety.

OTHER OUTCOMES:
Change in Behavioral Activation as Assessed by Behavioral Activation for Depression Scale - Short Form (BADS-SF) | Every week during the trial from baseline to post-intervention (week 0, 1, 2, 3, and 4)
  The level of behavioral activation among participants will be tracked through the course of treatment using BADS-SF. Participants will fill the BDS-SF every week at the treatment scheduled time. BADS-SF consists of 9 items with response on each item ranging from 0 to 6. The score of the BADS-SF will range from 0 to 54 with higher score indicating higher activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Puskesmas (Primary Healthcare Center), Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All IPD with supported informed consent that underlie results in a publication will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning at publication date with no end date
Access Criteria: The IPD and supporting information will be shared through Open Science Framework (OSF) Platform.